CLINICAL TRIAL: NCT01380275
Title: Docetaxel, Irinotecan, Recurrent, Refractory, Bone and Soft Tissue Sarcomas
Brief Title: Trial of Docetaxel and Irinotecan (DI) for Recurrent or Refractory Bone and Soft Tissue Sarcomas.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Byung-Kiu Park, Head of Center for Pediatric Oncology, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-08-322
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Sarcoma
Keywords: recurrent, refractory, bone, soft tissue, sarcomas
MeSH Terms: conditions — Sarcoma; Recurrence | interventions — Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel and Irinotecan (DI) (Experimental): Combination chemotherapy of Docetaxel and Irinotecan (DI) in recurrent or refractory bone and soft tissue sarcomas.
  Docetaxel and Irinotecan (DI) have different biologic targets, mode of action and mechanism of resistance. Preclinical studies have demonstrated an additive or synergistic effect of irinotecan and taxanes when used in combination in human.
  Docetaxel 100 mg/m2 mixed in D5W or N/S IV over 60 min: Day 1 Irinotecan 80 mg/m2 mixed in D5W IV over 90 min: Days 1 and 8 Therapy consists of 3-week cycles comprising weekly treatment for 2 weeks (docetaxel on D1 and irinotecan on D1 and D8) followed by 1-week rest, and will be continued in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel (Taxotere); Drug: Irinotecan

INTERVENTIONS:
Drug: Docetaxel (Taxotere) — This study : Docetaxel 100 mg/m2 mixed in D5W or N/S IV over 60 min: Day 1. Premedications : Dexamethasone 3 mg/m2 PO or IV 12 hours and 1 hour prior to docetaxel administration. A third dose of dexamethasone will be given 8 hours following docetaxel infusion. Patients should not be treated with docetaxel if they did not start the PO premedication the previous day. Parenteral pheniramine maleate may be given prior to docetaxel if patient has had a previous hypersensitivity to the agent. If used, pheniramine maleate (1 mg/kg IV) should be administered 30 minutes prior to infusion and every six hours thereafter, as needed.
  Other Names: Taxotere
Drug: Irinotecan — This study : Irinotecan 80 mg/m2 mixed in D5W IV over 90 min: Days 1 and 8. Premedications : Dexamethasone 3 mg/m2 PO or IV 12 hours and 1 hour prior to docetaxel administration. A third dose of dexamethasone will be given 8 hours following docetaxel infusion. Patients should not be treated with docetaxel if they did not start the PO premedication the previous day. Parenteral pheniramine maleate may be given prior to docetaxel if patient has had a previous hypersensitivity to the agent. If used, pheniramine maleate (1 mg/kg IV) should be administered 30 minutes prior to infusion and every six hours thereafter, as needed.

SUMMARY:
The purpose of this study is to estimate the control rate (CR,PR,SD) of docetaxel and irinotecan (DI) combination chemotherapy for recurrent or refractory bone and soft tissue sarcomas.Al so, this study is to evaluate the toxicity profile of Docetaxel and Irinotecan (DI) combination chemotherapy.

DETAILED DESCRIPTION:
Treatment setting:Hospitalization is preferred, but treatment on the outpatient base is allowed.

Regimen and premedication

1. Regimen Docetaxel 100 mg/m2 mixed in D5W or N/S IV over 60 min: Day 1 Irinotecan 80 mg/m2 mixed in D5W IV over 90 min: Days 1 and 8
2. Premedications Dexamethasone 3 mg/m2 PO or IV 12 hours and 1 hour prior to docetaxel administration. A third dose of dexamethasone will be given 8 hours following docetaxel infusion. Patients should not be treated with docetaxel if they did not start the PO premedication the previous day. Parenteral pheniramine maleate may be given prior to docetaxel if patient has had a previous hypersensitivity to the agent. If used, pheniramine maleate (1 mg/kg IV) should be administered 30 minutes prior to infusion and every six hours thereafter, as needed.

Treatment interval and overall treatment period : Therapy consists of 3-week cycles comprising weekly treatment for 2 weeks (docetaxel on D1 and irinotecan on D1 and D8) followed by 1-week rest, and will be continued in the absence of disease progression or unacceptable toxicity. Maximal number of cycles is twelve, however, additional cycles may be employed only when at least PR is maintained and patients want to take more.

Treatment modifications : Toxicity is evaluated according to common terminology criteria for adverse events v3.0 (CTCAE) of the National Cancer Institute.

Next cycle is to be delayed until ANC count on the starting day of scheduled treatment is at least 750/μL and platelet count is at least 75,000/μL, when full doses of irinotecan and docetaxel will be given. Next cycle is also delayed if diarrhea of grade 2 or higher (including moderate cramping) occurs on the day when the dose is due.

Irinotecan treatment of D8 will be delayed to D10 if grade 2 or higher non-hematological toxicity occurred on the day when the dose is due. Irinotecan scheduled at D8 will be omitted if diarrhea of grade 2 or higher occurred on the D10. Doses of docetaxel and irinotecan in the subsequent cycles are reduced by 20% for febrile grade 4 neutropenia (ANC<500/μL). Subsequent dose will be reduced by 20% for the recurrent toxicity. G-CSF is allowed if clinically indicated according to the ASCO guideline (22). Dose of docetaxel in the subsequent cycles are reduced by 20% for grade 2 neurologic toxicity/recurrent fluid retention, or any grade 3 non-hematologic toxicities, including hepatotoxicity, peripheral neuropathy, stomatitis, skin eruption, myalgia, cardiac events, or hypersensitivity. Subsequent dose will be reduced by 20% for the recurrent toxicity. In patients with grade 2 or higher fluid retention syndrome, prophylactic dexamethasone will be given by 6 mg/m2 bid for 3 days. Dose re-escalation after dose reduction is not permitted. Docetaxel and Irinotecan (DI) treatment will be discontinued in patients with grade 4 non-hematological toxicities at the discretion of investigators.

Dose modification schedule : Docetaxel and Irinotecan (DI) dose adjustment within a cycle will be made following the guidelines shown in Table 1 and 2 based on weekly WBC count and criteria for adverse events v3.0 (CTCAE).

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of rhabdomyosarcoma, liposarcoma, leiomyosarcoma, malignant fibrous histiocytoma, angiosarcoma, fibrosarcoma, malignant hemangiopericytoma, desmoplastic small round cell tumor, epitheloid sarcoma, clear cell sarcoma, synovial sarcoma, extraskeletal chondrosarcoma, alveolar soft part sarcoma, sarcoma not otherwise specified, malignant peripheral nerve sheath tumor, osteogenic sarcoma, Ewing's sarcoma/PPNET
2. One or more prior chemotherapy: Refractory tumors are defined as non-responsiveness to one or two regimens. In children less than 18 years, ifosfamide/carboplatin/etoposide (ICE) or VICE (vincristine + ICE) chemotherapy is recommended as a prior salvage regimen but is not mandatory.
3. Non-resectable recurrent or refractory rhabdomyosarcoma, liposarcoma, leiomyosarcoma, malignant fibrous histiocytoma, angiosarcoma, fibrosarcoma, malignant hemangiopericytoma, desmoplastic small round cell tumor, epitheloid sarcoma, clear cell sarcoma, synovial sarcoma, extraskeletal chondrosarcoma, alveolar soft part sarcoma, sarcoma not otherwise specified, malignant peripheral nerve sheath tumor, osteogenic sarcoma, Ewing's sarcoma/PPNET
4. Debulking surgery for non-resectable tumors is allowed when remained mass post-debulking is measurable enough to evaluate the response to DI.
5. Disease status must be that of measurable disease defined as:

   Lesions that can be accurately measured in at least one dimension with longest diameter >20mm using conventional techniques or >10mm with spiral CT scan.
6. Age less than 50 years
7. Predicted life expectancy of more than 8 weeks
8. Performance status: ECOG 0-2 or Karnofsky ≥ 50% for patients more than 10 years of age, and Lansky ≥ 50% for children equal or less than 10 years of age.
9. Adequate major organ function defined as; Hematopoietic function: ANC> 750/μL, platelet count>75,000/μL (If peripheral blood counts are inadequate due to bone marrow infiltration, then following a bone marrow biopsy to document disease, the patient will be eligible for study, but will be inevaluable for hematological toxicity. Patients with no increase in the infiltration of the marrow on follow-up marrow exams may receive further therapy with inadequate blood counts if they have recovered from all non-hematologic toxicities.) Hepatic function: bilirubin <1.5 mg/dL, AST/ALT levels <2.5 X UNL Renal function: creatinine <1.5 X UNL for age (Table 3) or GFR ≥ 50 ml/min/1.73m2
10. Patients must not receive any other anti-cancer agents or other investigational agents during the course of this investigation or within 3 weeks prior to study entry. At least 8 weeks must have elapsed since administration of extended radiotherapy or nitrosurea. Evaluable lesions must not have any radiotherapy within 8 weeks of the start of this protocol. Previously irradiated lesions that are used to evaluate tumor response must have shown evidence of an interim increase in size. For patients who have had stem cell transplant, they must have evidence of stable engraftment without the need for significant blood product support or cytokine therapy.
11. Patients and/or their parents or legal guardians should sign a written informed consent.

Exclusion Criteria:

1. Patients who have received either prior docetaxel or irinotecan.
2. Patients who are taking anticonvulsants.
3. Patients with uncontrolled infections.
4. Women of childbearing age must not be pregnant or lactating.
5. Inadequate cardiovascular function
6. Other malignancy within the past 3 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
7. Psychiatric disorder that would preclude compliance

Ages: 5 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-04; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
CT or MRI image of tumor | 2 cycles after chemotherapy (6 weeks, 1cycle = 3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Kiu Park, M.D.,Ph.D., Principal Investigator — Pediatric Oncology Branch, National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Yoon JH, Kwon MM, Park HJ, Park SY, Lim KY, Joo J, Park BK. A study of docetaxel and irinotecan in children and young adults with recurrent or refractory Ewing sarcoma family of tumors. BMC Cancer. 2014 Aug 28;14:622. doi: 10.1186/1471-2407-14-622. PMID 25164234